CLINICAL TRIAL: NCT04254263
Title: Adjuvant Trastuzumab Plus Pyrotinib for Residual Invasive HER2-positive Breast Cancer After Neoadjuvant Chemotherapy Plus Anti-HER2 Target Therapy
Brief Title: Adjuvant Study of Pyrotinib in HER-2 Positive Breast Cancer
Acronym: ATP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2019-070
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Breast Cancer
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyrotinib (Experimental): pyrotinib 400 mg, orally once daily for one year
  Interventions: Drug: pyrotinib
- No Pyrotinib (No Intervention): Observation follow-up

INTERVENTIONS:
Drug: pyrotinib — pyrotinib 400 mg, orally once daily for one year
  Arms: Pyrotinib

SUMMARY:
This is a prospective, randomised, multicenter, no placebo-controlled, open label study for evaluating the efficacy and safety of pyrotinib in women with residual invasive HER2-positive breast cancer after neoadjuvant chemotherapy plus anti-HER2 target therapy. The main purpose is to investigate whether pyrotinib can further reduce the risk of recurrence from previously diagnosed HER-2 positive breast cancer based on the 1-year trastuzumab standard adjuvant treatment with or without pertuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Female, Aged ≥18 and ≤70 years;
* Histologically confirmed invasive HER2 positive breast cancer, early disease(Stage ⅡA-Ⅲ) ;
* Completed neoadjuvant therapy, including chemotherapy and trastuzumab;
* Residual invasive disease was detected pathologically in the surgical specimen of the breast or axillary lymph nodes after completion of neoadjuvant chemotherapy;
* Been or being treated for early breast cancer with standard of care duration of trastuzumab;
* Adjuvant treatment regimen needs to be determined before randomization;
* Duration from Random time to the last use of trastuzumab≤1 year.
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1;
* Required laboratory values including following parameters:ANC: ≥ 1.5 x 109/L; Platelet count: ≥ 100 x 109/L; Hemoglobin: ≥ 9.0 g/dL; Total bilirubin: ≤ 1.5 x upper limit of normal, ULN; ALT and AST: ≤ 1.5 x ULN; BUN and creatine clearance rate: ≥ 50 mL/min; LVEF: ≥ 50%; QTcF: < 470 ms
* Signed informed consent form (ICF) .

Exclusion Criteria:

* Metastatic disease (Stage IV) ;
* Gross residual disease remaining after mastectomy or positive margins after breast-conserving surgery;
* Progressive disease during neoadjuvant therapy;
* Subjects that are unable to swallow tablets, or dysfunction of gastrointestinal absorption;
* Treated or treating with anti-HER2 TKI, including but not limited to pyrotinib, lapatinib and neratinib.
* Less than 4 weeks from the last clinical trial;
* History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation;
* Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial;
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test;Female patients of childbearing age that are reluctant to take effective contraceptive measures throughout the trial period;
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (iDFS) | From randomization until time of event up to 2 years.
  Invasive disease-free survival time is defined as the time from date of randomization until the first invasive disease recurrence of the following events: invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, distant recurrence and death from any cause.

SECONDARY OUTCOMES:
Disease-free Survival (DFS) | From randomization until time of event up to 2 years
  Disease-free survival time is defined as the time from date of randomization until the first disease recurrence of the following events: invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, non-breast primary invasive cancer, ductal carcinoma in situ(DCIS),or distant recurrence and death from any cause
Overall Survival (OS) | From randomization until time of event up to 2 years
  Overall survival is defined as the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Lu, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided